CLINICAL TRIAL: NCT00296673
Title: Reactive Neuromuscular Training Effects on Side Bridge Endurance Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LCC-06-01
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Balance
Keywords: Rehabilitation, Side Bridge test, Muscular endurance

INTERVENTIONS:
Device: Rehabilitation device

SUMMARY:
The purpose of this study is to determine the effects of reactive neuromuscular training on muscular endurance test.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants with no history of balance problems, ages 20 - 40.

Exclusion Criteria:

1. Lower extremity injury, surgery, visual, or vestibular condition that would effect balance?
2. Unstable joints of the lower extremity infections, injuries or other malignancies affecting the lower extremity?

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Study Completion 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Dennis E. Enix, DC, Principal Investigator — Logan College of Chiropractic; Rodger E. Tepe, PhD, Study Director — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States

REFERENCES:
- [Background] Visser JE, Bloem BR. Role of the basal ganglia in balance control. Neural Plast. 2005;12(2-3):161-74; discussion 263-72. doi: 10.1155/NP.2005.161. PMID 16097484
- [Background] Delecluse C, Roelants M, Verschueren S. Strength increase after whole-body vibration compared with resistance training. Med Sci Sports Exerc. 2003 Jun;35(6):1033-41. doi: 10.1249/01.MSS.0000069752.96438.B0. PMID 12783053
- [Background] Jemmett RS, Macdonald DA, Agur AM. Anatomical relationships between selected segmental muscles of the lumbar spine in the context of multi-planar segmental motion: a preliminary investigation. Man Ther. 2004 Nov;9(4):203-10. doi: 10.1016/j.math.2004.07.006. PMID 15522645
- [Background] Chiang J, Potvin JR. The in vivo dynamic response of the human spine to rapid lateral bend perturbation: effects of preload and step input magnitude. Spine (Phila Pa 1976). 2001 Jul 1;26(13):1457-64. doi: 10.1097/00007632-200107010-00016. PMID 11458151
- [Background] Shiavi RG, Champion SA, Freeman FR, Bugel HJ. Efficacy of myofeedback therapy in regaining control of lower extremity musculature following stroke. Am J Phys Med. 1979 Aug;58(4):185-94. PMID 464030